CLINICAL TRIAL: NCT04919265
Title: Breastmilk, Infant Gut Microbiome and the Impact on Infant Health: a Prospective Mother-Infant Cohort Study in Malaysia and China
Brief Title: Mother-Infant Cohort Study in Malaysia and China
Status: Recruiting | Type: Observational
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: Guilin University of Technology, China (Unknown); National Engineering Center of Dairy for Maternal and Child Health, Beijing (Unknown)
Responsible Party: Principal Investigator, Gan Wan Ying, Assoc. Prof. Dr., Universiti Putra Malaysia
Other Study IDs: SANYUANUPM
Record Dates: First submitted 2021-05-19; First posted 2021-06-09 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Gut Microbiota; Gastrointestinal Symptoms; Temperament; Eczema; Asthma; Breast Milk Collection
Keywords: Gut microbiota; Mother-infant cohort study; Breastmilk
MeSH Terms: conditions — Eczema; Asthma; Breast Milk Expression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During pregnancy: maternal blood. At delivery: mother's milk. During infancy: Mother's saliva, blood, milk, feces, and urine as well as baby's saliva, blood, feces, and urine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Mother and Infant: The cohort will be followed for 2 years with 8 follow-up measurement points of the infants until the age of 1 year.
  Interventions: Other: No intervention - mother-infant cohort study

INTERVENTIONS:
Other: No intervention - mother-infant cohort study — There are no interventions because it is a mother-infant cohort study

SUMMARY:
This mother-infant cohort study aims to determine the geographic differences in the microbial profiles in breast milk from mothers living in Malaysia and China that are potentially important determinants of infant development. It also aims to determine the impact of gut microbiome on infant health (temperament, gastrointestinal symptoms, eczema symptoms, and asthma symptoms).

DETAILED DESCRIPTION:
Gut microbiota plays a critical role in children's developmental pathways especially in the first 1000 days of life. A number of pre- and post-natal factors were known to affect gut microbiota in infants during their first year of life including mode of delivery, infant feeding practices, dietary intake, and human milk composition. However, there is no mother-infant cohort study comparing gut microbiota profile and breastmilk composition of mothers living in Malaysia and China. Recent studies showed that gut microbiota was associated with infant health including temperament, gastrointestinal disorders, eczema, and asthma. However, little is known about the gut microbiome and the factors that contribute to microbial variation in the gut of South East Asian children. Increased awareness on the importance of gut health helps establish pre-natal and post-natal factors that promote healthy development and functioning of immune system, gastrointestinal health, and metabolism in infants.

This study is a prospective cohort study involving pregnant women in the first trimester of pregnancy. Data will be collected from the eligible pregnant women during their first trimester (8-12 weeks of gestation), second trimester (24 weeks of gestation), third trimester (34 weeks of gestation) and follow-up infants and mothers postnatally after birth (1-5 days after delivery), at 10-15 days, 1 month, 4 months and 12 months of age with a total of 8 follow-ups of mother-infant biological samples and related research data.

Mothers will be interviewed on socio-demographic background and information on pre-natal and post-natal factors such as obstetric history, exposure to antibiotics/prebiotics/probiotics/ paracetamol, pre-pregnancy body BMI, gestational weight gain, GDM, physical activity, food security, smoking during pregnancy/second-hand exposure, dietary intake, stress during pregnancy, home settings, pet keeping, and post-natal depression. Mothers will also be interviewed on their infants' sex, birth order, gestational age, mode of delivery, body weight, length, and head circumferences, second hand smoke exposure, exposure to antibiotics/prebiotics/probiotics/paracetamol, infant feeding practices, dietary intake, and dietary diversity. Anthropometric measurements of mothers and infants will be conducted at every visit. Blood, fecal, saliva, and urine samples of mothers and infants will also be collected. All bio-specimens are stored at -80°C until they are transported to National Engineering Center of Dairy for Maternal and Child Health, Beijing, China for further analysis.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged between 18 and 45 years old
* Pregnant women who attend the antenatal check-up at the selected clinics/hospitals
* Pregnant women with the gestational age of less than 12 weeks
* Pregnant women who plan to attend post-natal check-ups for at least one year at the same clinic/hospital

Exclusion Criteria:

* Pregnant women who are diagnosed with immune deficiency
* Pregnant women who have a multiple pregnancy and preterm delivery (<37 weeks)
* Pregnant women who plan to move out of the study area in the next one year
* Pregnant women with fetal/newborn with congenital abnormalities

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women in the first trimester of pregnancy will be recruited.
Study Population: Pregnant women in their first trimester of pregnancy (gestational age of less than 12 weeks) who visit the selected health clinics/hospitals will be invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-06-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Breastmilk microbiome | from birth to 12 months
  Breastmilk microbiota composition is determined by using 16S rRNA gene sequencing
Gut microbiome | from birth to 12 months
  Gut microbiome diversity profile is analysed from the stool by using qPCR and sequencing approaches analysis

SECONDARY OUTCOMES:
Temperament | 12 months
  Infant temperament is assessed using Revised Infant Behavior Questionnaire (IBQ-R) (Gartstein & Rothbart, 2003). It consists of 91 items with 14 subscales, including activity level, distress to limitations, high pleasure, low pleasure, soothability, falling reactivity, cuddliness, perceptual sensitivity, sadness, approach, and vocal reactivity. Mothers are requested to report their infants' behaviors during specific events in the past week using a 7-point scale, ranging from 1 (never) to 7 (always). Total scores of each dimensions range from 1 to 7, with a higher dimension score indicates higher tendency towards the dimension.
Gastrointestinal symptoms | from birth to 12 months
  Mothers are required to complete the Rome IV Diagnostic Questionnaire for Pediatric Functional Gastrointestinal Disorders-Toddler (R4PDQ-toddler) about their child's GI symptoms (Van Tilburg et al., 2016). Those who fulfill criteria for the last 3 months with symptom onset at least 6 months prior to diagnosis are considered as having gastrointestinal problem.
Eczema symptoms | from birth to 12 months
  The presence of eczema in infants will be determined based on five questions of the UK Working Party's Diagnostic Criteria for Atopic Dermatitis (Williams et al., 1994) with response options "yes" or "no". Total scores range from 0 to 5. Higher score indicates presence of eczema. Eczema in infants will be identified by the presence of an itchy skin condition plus 2 or more of the followings: (1) History of involvement of skin creases such as folds of elbows, behind the knees, fronts of ankles cheeks, or around the neck, (2) A history of atopic disease in a first-degree relative, (3) A history of a general dry skin, and (4) Visible flexural eczema.
Asthma symptoms | from birth to 12 months
  The Asthma Predictive Index (API) (Castro-Rodríguez et al., 2000) is used to determine the likelihood of infants who may develop asthma. A positive API score requires recurrent episodes of wheezing during the first 3 years of life and 1 of 2 major criteria (physician-diagnosed eczema or parental asthma) or 2 of 3 minor criteria (physician-diagnosis allergic rhinitis, wheezing without colds, or peripheral eosinophilia ≥4%). A loose index (<3 episodes/y and 1 of the major or 2 of the minor criteria) and a stringent index (≥3 episodes/year and 1 of the major or 2 of the minor criteria) are available.
Infant diet | from birth to 12 months
  breastfeeding duration in months
Infant height | from birth to 12 months
  height in cm
Infant weight | from birth to 12 months
  weight in kg

CONTACTS AND LOCATIONS:
Overall Officials: Wan Ying Gan, PhD, Principal Investigator — Universiti Putra Malaysia; Tie Min Jiang, Principal Investigator — Guilin University of Technology; Li Jun Chen, PhD, Study Director — Beijing Sanyuan Foods Co Ltd
Locations (1):
- Private hospital, Kajang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gartstein MA, Rothbart MK. Studying infant temperament via the Revised Infant Behavior Questionnaire. Infant Behavior and Development. 2003;26(1):64-86. https://doi.org/10.1016/S0163-6383(02)00169-8
- [Background] van Tilburg MA, Rouster A, Silver D, Pellegrini G, Gao J, Hyman PE. Development and Validation of a Rome III Functional Gastrointestinal Disorders Questionnaire for Infants and Toddlers. J Pediatr Gastroenterol Nutr. 2016 Mar;62(3):384-6. doi: 10.1097/MPG.0000000000000962. PMID 26308319
- [Background] Williams HC, Burney PG, Hay RJ, Archer CB, Shipley MJ, Hunter JJ, Bingham EA, Finlay AY, Pembroke AC, Graham-Brown RA, et al. The U.K. Working Party's Diagnostic Criteria for Atopic Dermatitis. I. Derivation of a minimum set of discriminators for atopic dermatitis. Br J Dermatol. 1994 Sep;131(3):383-96. doi: 10.1111/j.1365-2133.1994.tb08530.x. PMID 7918015
- [Background] Castro-Rodriguez JA, Holberg CJ, Wright AL, Martinez FD. A clinical index to define risk of asthma in young children with recurrent wheezing. Am J Respir Crit Care Med. 2000 Oct;162(4 Pt 1):1403-6. doi: 10.1164/ajrccm.162.4.9912111. PMID 11029352
- [Derived] Eow SY, Gan WY, Jiang T, Loh SP, Lee LJ, Chin YS, Than LTL, How KN, Thong PL, Liu Y, Zhao J, Chen L. MYBIOTA: A birth cohort on maternal and infant microbiota and its impact on infant health in Malaysia. Front Nutr. 2022 Sep 27;9:994607. doi: 10.3389/fnut.2022.994607. eCollection 2022. PMID 36238465